CLINICAL TRIAL: NCT02727530
Title: The Effects of Visceral Manual Therapy on Infant Colic Symptoms. A Controlled Clinical Trial
Brief Title: The Effectiveness of the Manual Therapy on Infant Colic (MT-IF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Raquel Chillón Martínez, PhD, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USeville-RMartinez
Record Dates: First submitted 2016-03-29; First posted 2016-04-04 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-04

CONDITIONS: Infant Colic
Keywords: Infant Colic; Manual Therapy; Effectiveness
MeSH Terms: conditions — Colic | interventions — Counseling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- GROUP RECEIVING VISCERAL MANUAL THERAPY-ADVICES (Experimental): Subjects will receive 2 manual therapy sessions and advices.
  Interventions: Other: VISCERAL MANUAL THERAPY-ADVICES; Other: ADVICES
- GROUP RECEIVING ADVICES (Experimental): Subjects will receive advices.
  Interventions: Other: ADVICES

INTERVENTIONS:
Other: VISCERAL MANUAL THERAPY-ADVICES — The subjects of this group will receive an amount of two sessions of visceral manual therapy that will be applied within two weeks. In the first session will be applied procedures in the most superficial body structures. And, in the second session will be applied procedures in the most deep body structures.
  Arms: GROUP RECEIVING VISCERAL MANUAL THERAPY-ADVICES
Other: ADVICES — Advices for parents to improve the management of infant colic

SUMMARY:
The main goal of this study is to get to know if applying manual therapy will reduce the infant colic symptoms for to improve quality of life of babies and parents.

DETAILED DESCRIPTION:
Background:

Infant colic is one of the most common disorders in the first year of baby´s life. It is estimated to affect between 10 to 40 % of healthy born children in their first year of life. To determine the effectiveness of a protocol manual therapy in the treatment of colic, using the Infant Colic Severity Questionnaire, we analyzed two intervention groups: experimental in which children received the protocol manual therapy and counseling to parents and the Control group, in which parents received advice only.

Objectives:

To assess the effectiveness of visceral manual therapy to improve the symptoms on infant colic.

ELIGIBILITY:
Inclusion Criteria:

* Infants with medical diagnostic of colic following Wessel criteria.

Exclusion Criteria:

* Infant's parents without full capacity to answer the survey questions, such as the existence of intellectual disability.
* Babies with neurological disorders such epilepsy, meningitis, encephalitis, cerebral palsy, spina bifida, hydrocephalus, encephalopathy, Arnold Chiari malformation, syringomyelia and Huntington's disease.
* Babies with digestive disorders, such Crohn's disease, irritable bowel syndrome, peritonitis, intestinal malabsorption, hepatitis, diverticular bowel disease, esophagitis, Intussusception and Ulcerative Colitis.
* Babies with congenital diseases such Angelmen syndrome, Down syndrome, cystic fibrosis, haemophilia, Klinefelter syndrome, Neurofibromatosis, Patau syndrome and Tay Sachs syndrome.
* Babies with traumatology - orthopedic pathologies such idiopathic scoliosis, spondylolisthesis, Perthes disease, Meyer dysplasia, Marfan syndrome, Morquio syndrome and congenital hip dislocation.
* Babies with dermatological diseases such Atopic dermatitis, staphylococcal scalded skin syndrome, psoriasis, urticaria and disorders of skin pigmentation.
* Babies who are subjected to drug treatments that are not specific to the treatment of colic.

Ages: 1 Day to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from parents-reported infant colic severity at 3 weeks | At the start of the study and one week after the second session (three weeks after the start of the study)
  Evaluated by the infant colic severity scale

SECONDARY OUTCOMES:
Change from parents-reported infant cry at 3 weeks | At the start of the study and one week after the second session (three weeks after the start of the study)
  Evaluated by cry-related items of the infant colic severity scale

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo de Investigación Área de Fisioterapia CTS 305 - Universidad de Sevilla, Seville, Sevilla, Spain

REFERENCES:
- [Result] WESSEL MA, COBB JC, JACKSON EB, HARRIS GS Jr, DETWILER AC. Paroxysmal fussing in infancy, sometimes called colic. Pediatrics. 1954 Nov;14(5):421-35. No abstract available. PMID 13214956
- [Result] Wurmser H, Laubereau B, Hermann M, Papousek M, von Kries R. Excessive infant crying: often not confined to the first 3 months of age. Early Hum Dev. 2001 Aug;64(1):1-6. doi: 10.1016/s0378-3782(01)00166-9. PMID 11408103
- [Result] Ernst E. Chiropractic spinal manipulation for infant colic: a systematic review of randomised clinical trials. Int J Clin Pract. 2009 Sep;63(9):1351-3. doi: 10.1111/j.1742-1241.2009.02133.x. PMID 19691620
- [Result] Olafsdottir E, Forshei S, Fluge G, Markestad T. Randomised controlled trial of infantile colic treated with chiropractic spinal manipulation. Arch Dis Child. 2001 Feb;84(2):138-41. doi: 10.1136/adc.84.2.138. PMID 11159288
- [Result] Reinthal M, Lund I, Ullman D, Lundeberg T. Gastrointestinal symptoms of infantile colic and their change after light needling of acupuncture: a case series study of 913 infants. Chin Med. 2011 Aug 11;6:28. doi: 10.1186/1749-8546-6-28. PMID 21835014
- [Result] Skjeie H, Skonnord T, Fetveit A, Brekke M. Acupuncture for infantile colic: a blinding-validated, randomized controlled multicentre trial in general practice. Scand J Prim Health Care. 2013 Dec;31(4):190-6. doi: 10.3109/02813432.2013.862915. Epub 2013 Nov 15. PMID 24228748
- [Result] Larsen JH. Infants' colic and belly massage. Practitioner. 1990 Apr 22;234(1487):396-7. No abstract available. PMID 2367295